CLINICAL TRIAL: NCT04484974
Title: A Randomized, Two Condition, Crossover Trial Assessing Appetite, Energy Metabolism, Blood Biomarker and ad Libitum Food Intake Responses to a Mid-morning Pecan Snack vs. an Equicaloric High Carbohydrate Savory Snack in Healthy Volunteers With Overweight/Obesity
Brief Title: Effects of Pecan Nut Snacks v Equicaloric Snacks on Appetite, Food Intake, Metabolism, Hormones and Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Pecan Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-0048
Record Dates: First submitted 2020-06-26; First posted 2020-07-24 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Overweight and Obesity
Keywords: Pecans; appetite; hormones; food intake
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: Randomized, two period crossover with two treatment conditions
Masking Description: The two treatments are pecan nuts or tortilla chips as snacks, therefore masking of treatment conditions is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecan snack condition (Experimental): In this crossover condition, a mid morning snack consisting of 250 kcal of lightly salted roasted pecan nuts will be administered.
  Interventions: Other: Pecan snack
- Tortilla chip snack condition (Active Comparator): In this crossover condition, a mid morning snack consisting of 250 kcal of lightly salted pretzels will be administered.
  Interventions: Other: Tortilla chip snack

INTERVENTIONS:
Other: Pecan snack — Under this condition, each participant will consume a mid morning snack of pecans followed by an ad libitum lunch.
  Arms: Pecan snack condition
Other: Tortilla chip snack — Under this condition, each participant will consume a mid morning snack consisting of an iso-caloric (equal to the pecan snack) snack of tortilla chips followed by an ad libitum lunch.
  Arms: Tortilla chip snack condition

SUMMARY:
This is a within-subjects crossover study that examines subjective appetite, food intake, hormone and metabolic responses to consumption of mid morning snacks of pecan nuts as compared to an iso-caloric amount of tortilla chips. Pecans are high in fat and calories and low in carbohydrate by weight, while tortilla chips are mostly carbohydrate and essentially devoid of fat. These two very different nutrient profiles should elicit different metabolic and biomarker responses. The study aims to determine whether these treatments also elicit different subjective appetite and food intake responses. Participants will be healthy volunteers with overweight and obesity, a population that may be seeking healthy snacking options that are satisfying and satiating.

DETAILED DESCRIPTION:
This is a randomized, two condition, crossover study in healthy individuals with overweight and obesity examining the effect of a mid-morning snack of pecans vs. a low fat savory snack on appetite, energy expenditure, blood biomarkers of appetite and metabolism and ad libitum food intake at lunch. Twenty-four participants will be enrolled and studied on two test days with at least one week washout in between. On test days, participants will have baseline measures of appetite (by Visual Analogue Scale (VAS)), blood hormones and substrates, and energy expenditure and fuel oxidation (Resting Metabolic Rate (RMR), by indirect calorimetry) taken just prior to consuming a standardized 300 kcal breakfast. VAS measures will be taken at 20, 30, 60, 90 and 120 min following the meal and RMR will be measured for 20 min after eating. A mid-morning snack of either 250 kcal of pecans or lightly salted tortilla chips will be consumed and VAS and blood measures will be taken at 20, 30, 60, 90 and 120 min following the snack and RMR will be measured for 20 min after eating. Participants will be given an ad libitum lunch meal and VAS and blood measures will be taken at 20, 30, 60, 90 and 120 min following the lunch and RMR will be measured for 20 min after eating. Blood will be analyzed for glucose, insulin, free fatty acids, triglycerides, ghrelin, leptin, PYY, and GLP-1. Two hypotheses will be examined: 1. pecans will provoke greater feelings of fullness and reduced hunger after the snack and lunch meal consumption (on either a calorie per calorie or volume basis) as compared to the tortilla chip snack, and 2. the pecan snack will provoke greater responses of satiety hormones compared to tortilla chips. Post-snack and lunch energy expenditure and fat oxidation will also be compared between treatments as an exploratory aim.

ELIGIBILITY:
Inclusion Criteria:

1. 35 adult men and women
2. all ethnic groups
3. ages 20-50,
4. BMI 27-35,
5. habitually eat breakfast,
6. willing to eat the test snacks and other foods offered,
7. weight stable for the last 6 months
8. willing to consent and adhere to the test procedures and schedule

Exclusion Criteria:

1. nut allergies,
2. uncontrolled thyroid disorders,
3. diabetes mellitus,
4. eating disorders,
5. pregnant, or planning to become pregnant during the study,
6. lactating,
7. uncontrolled hypertension,
8. active dieting
9. intensive physical activity training regimen (>300 min/wk exercise),
10. medical history or current medication that may affect study outcomes per study PI discretion
11. consuming pecans on a regular basis
12. unable to lie still with a clear hood over their head for the measurement of energy expenditure

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline (before snack consumption) to 120 minutes in subjective appetite response to pecan or pretzel snack using visual analog assessment | Baseline (prior to mid-morning snack consumption) to 120 minutes after snack consumption at 20, 30, 60, 90 and 120 minutes following consumption.
  Subjective appetite will be assessed using a visual analog scale. Subjective feelings will be rated on a 100 mm horizontal line preceded by the questions: "How hungry are you right now?" and anchored on the left by "not at all hungry" and by "extremely hungry" on the right; Fullness will be queried by "How full do you feel right now?" anchored by "not at all..." and "extremely..."; Desire to eat will be queried by, "How strong is your desire to eat right now?" anchored by anchored by "not at all..." and "extreme...; and prospective consumption will be queried by, "how much food do you think you can you eat right now" with anchors of "not (much) at all" to "extremely/an extreme amount".
Change from baseline (prior to lunch) to 120 minutes in subjective appetite response to lunch meal using visual analog assessment | Prior to lunch consumption and at 20, 30, 60, 90 and 120 minutes following consumption.
  Subjective appetite will be assessed using a visual analog scale. Subjective feelings will be rated on a 100 mm horizontal line preceded by the questions: "How hungry are you right now?" and anchored on the left by "not at all hungry" and by "extremely hungry" on the right; Fullness will be queried by "How full do you feel right now?" anchored by "not at all..." and "extremely..."; Desire to eat will be queried by, "How strong is your desire to eat right now?" anchored by anchored by "not at all..." and "extreme...; and prospective consumption will be queried by, "how much food do you think you can you eat right now" with anchors of "not (much) at all" to "extremely/an extreme amount".
Energy intake response to pecan or pretzel snack using weighed food intake measures | 30 minutes allowed for completion of the lunch meal
  Energy intake at ad libitum lunch meal consisting of a variety of different foods offering approximately 1400 of kilocalories of energy having an overall composition of approximately 15% protein, 55% carbohydrate and 30% fat. Twelve ounces of water will be provided as the beverage. Energy intake will be calculated from the weight of each food consumed and the published nutrient composition of the foods. Linear mixed effects model will be used to test the difference in energy intake between two experimental conditions.
Change from baseline (prior to snack consumption) to 120 minutes in serum glucose following pecan or pretzel snack consumption. | Baseline (prior to snack) to 120 minutes at intervals of 20, 30, 60, 90 and 120 minutes.
  Serum glucose by enzymatic method.
Change from baseline (prior to lunch consumption) to 120 minutes in serum glucose following lunch consumption. | Prior to lunch and at intervals of 20, 30, 60, 90 and 120 minutes after lunch consumption.
  Serum glucose by enzymatic method.
Change from baseline (prior to snack consumption) to 120 minutes in serum insulin following pecan or pretzel snack consumption. | Prior to snack and at intervals of 20, 30, 60, 90 and 120 minutes after snack consumption.
  Serum insulin by radio-immunoassay.
Change from baseline (prior to lunch consumption) to 120 minutes in serum insulin following lunch consumption. | Prior to lunch and at intervals of 20, 30, 60, 90 and 120 minutes after lunch consumption.
  Serum insulin by radio-immunoassay.
Change from baseline (prior to snack consumption) to 120 minutes in serum triglycerides following pecan or pretzel snack consumption. | Prior to snack and at intervals of 20, 30, 60, 90 and 120 minutes after snack consumption.
  Serum triglycerides by enzymatic assay.
Change from baseline (prior to lunch consumption) to 120 minutes in serum triglycerides following lunch consumption. | Prior to lunch and at intervals of 20, 30, 60, 90 and 120 minutes after lunch consumption.
  Serum triglycerides by enzymatic assay.
Change from baseline (prior to snack consumption) to 120 minutes in serum free fatty acids following snack consumption. | Prior to mid-morning snack and at intervals of 20, 30, 60, 90 and 120 minutes after snack consumption.
  Serum free fatty acids by enzymatic assay.
Change from baseline (prior to lunch consumption) to 120 minutes in serum free fatty acids following lunch consumption. | Prior to lunch and at intervals of 20, 30, 60, 90 and 120 minutes after lunch consumption.
  Serum free fatty acids by enzymatic assay.
Change from baseline (prior to snack consumption) to 120 minutes in serum ghrelin following snack consumption. | Prior to mid-morning snack and at intervals of 20, 30, 60, 90 and 120 minutes after snack consumption.
  Serum ghrelin by radio-immunoassay
Change from baseline (prior to lunch consumption) to 120 minutes in serum ghrelin following lunch consumption. | Prior to lunch and at intervals of 20, 30, 60, 90 and 120 minutes after lunch consumption.
  Serum ghrelin by radio-immunoassay
Change from baseline (prior to snack consumption) to 120 minutes in serum peptide YY following snack consumption. | Prior to snack and at intervals of 20, 30, 60, 90 and 120 minutes after snack consumption.
  Serum peptide YY (PYY) by radio-immunoassay
Change from baseline (prior to lunch consumption) to 120 minutes in serum peptide YY following lunch consumption. | Prior to lunch and at intervals of 20, 30, 60, 90 and 120 minutes after lunch consumption.
  Serum peptide YY (PYY) by radio-immunoassay
Change from baseline (prior to snack consumption) to 120 minutes in serum glucagon like peptide-1 following snack consumption. | Prior to snack and at intervals of 20, 30, 60, 90 and 120 minutes after snack consumption.
  Serum glucagon like peptide-1 (GLP-1) by enzyme immunoassay
Change from baseline (prior to lunch consumption) to 120 minutes in serum glucagon like peptide-1 following lunch consumption. | Prior to lunch and at intervals of 20, 30, 60, 90 and 120 minutes after lunch consumption.
  Serum glucagon like peptide-1 (GLP-1) by enzyme immunoassay
Change in serum leptin from baseline to 120 minutes following snack consumption | Baseline (prior to breakfast) and at 120 minutes following mid-morning snack consumption.
  Serum leptin by immunoassay.

SECONDARY OUTCOMES:
Change from baseline in energy expenditure post snack | Resting energy expenditure will be measured for 20 minutes after snack consumption.
  Post snack resting energy expenditure will be measured using hood indirect calorimetry. Energy expenditure will be measured using standard indirect calorimetry with the ventilated hood technique (Parvo Medics Truemax 2400, Salt Lake City, UT).
Change from baseline in energy expenditure post lunch | Resting energy expenditure will be measured for 20 minutes after lunch consumption.
  Post lunch resting energy expenditure will be measured using hood indirect calorimetry. Energy expenditure will be measured using standard indirect calorimetry with the ventilated hood technique (Parvo Medics Truemax 2400, Salt Lake City, UT).

CONTACTS AND LOCATIONS:
Overall Officials: John C Peters, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Health and Wellness Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No